CLINICAL TRIAL: NCT02306850
Title: Phase 2B Single-site, Open-label, Nonrandomized Study Evaluating the Efficacy of Neoadjuvant Pembrolizumab for Unresectable Stage III and Unresectable Stage IV Melanoma
Brief Title: Neoadjuvant Pembrolizumab for Unresectable Stage III and Unresectable Stage IV Melanoma
Acronym: NeoPembroMel
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, John Richart, M.D., Associate Professor, Dept. of Internal Medicine, Hematology and Oncology, St. Louis University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SLU IRB 25007; 51604 (Other: Merck)
Record Dates: First submitted 2014-12-01; First posted 2014-12-03 (Estimated); Results first posted 2019-06-20 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Unresectable Malignant Neoplasm; Melanoma; Metastatic Melanoma; Stage IV Melanoma; Stage III Melanoma
Keywords: immunotherapy; PD-1 inhibitor; programmed death 1 inhibitor; neoadjuvant; pembrolizumab; MK-3475
MeSH Terms: conditions — Melanoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pembrolizumab (Experimental): Open-label non-randomized trial. All subjects will receive active drug (pembrolizumab).
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — At the Treatment Initiation Visit (Baseline/Day 1), subjects will begin treatment with IV pembrolizumab 200 mg infusions every 3 weeks. As in previous pembrolizumab trials, eligible subjects will receive at least 24 weeks of therapy and may receive up to 2 years of pembrolizumab therapy depending on response to treatment.
  Other Names: Keytruda; MK-3475

SUMMARY:
This study is being done to see if using the study drug, pembrolizumab, can shrink down melanoma tumors enough so that they will be small enough to cut out, so that there will be no cancer left in the body.

Eligible participants include those who have not received any systemic melanoma therapies (i.e. participants do not have to fail ipilimumab or BRAF inhibitor) and those who have failed all available systemic options (if the participant meets other inclusion / exclusion criteria).

DETAILED DESCRIPTION:
This study is being done to see if using the study drug, pembrolizumab, can shrink down melanoma tumors enough so that they will be small enough to cut out, so that there will be no cancer left in the body.

Eligible participants include those who have not received any systemic melanoma therapies (i.e. participants do not have to fail ipilimumab or BRAF inhibitor) and those who have failed all available systemic options (if the participant meets other inclusion / exclusion criteria).

For most melanoma cases, surgery is the recommended treatment. Until recently surgery was not used for patients with advanced melanoma (melanoma that has spread to lymph nodes or melanoma that has spread to other organs like the lung, liver, brain) because it was thought that surgery wouldn't help patients live longer when the melanoma tumors had spread beyond the skin. Recent studies have shown that patients with advanced melanoma who have surgery as one of their treatments may live longer than patients who only have systemic therapy (IV drugs or pills) and do not have surgery at all.

Unfortunately, when patients with advanced melanoma come to the doctor, surgery is not a good choice for most patients because they have 'unresectable' melanoma. 'Unresectable' melanoma means they have melanoma tumors in the body that are too big or too close to important parts in the body (like big blood vessels) to be cut out safely. We are studying if we can use a drug to shrink tumors down to make them small enough to cut out; this is called a "neoadjuvant" approach to treating melanoma. By removing all of the cancer from body by using the combination of drug and surgery, we think this could help people live longer.

Pembrolizumab is a drug that is given in the veins and can make the immune system stronger so that it can fight cancer cells. Pembrolizumab is in the class of drugs called immunotherapy.

Immunotherapy uses parts of a person's immune system to fight the disease. Pembrolizumab is designed to restore the natural ability of the immune system to recognize and target melanoma cells to be attacked. In addition to possibly shrinking tumors, it may change your immune system so that it can fight melanoma in the future.

We are also trying to learn more about how pembrolizumab works in the body. In this study, we will look at the skin, blood, and bone marrow to see if we can see any signs to tell doctors whether pembrolizumab is working or tell us which patients it may work on.

ELIGIBILITY:
Inclusion Criteria:

1. Be able to provide written informed consent.
2. Be 18 years old at time of consent.
3. Have measurable disease by RECIST 1.1.
4. Has a diagnosis of unresectable Stage III or Stage IV melanoma with anatomic site(s) of metastasis that could be amenable to curative resection if the site(s) decreased in size by up to 50% (at the investigators' discretion).
5. Have provided tissue sample of a tumor lesion.
6. Have an ECOG Performance status 0 or 1.
7. Demonstrate adequate organ function according to pre-defined criteria
8. Females of childbearing potential should have a negative pregnancy test within 72 hours prior to receiving the first dose.
9. Females of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity during the study through 120 days after last dose. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.

10 . Males should agree to use an adequate method of contraception starting with the first dose of therapy through 120 days after last dose.

Exclusion Criteria:

1. Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment.
2. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of treatment.
3. Has had a prior monoclonal antibody within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered > 4 weeks earlier.
4. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.
5. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell and squamous cell skin cancers, or in situ cervical cancer.
6. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging 4 weeks prior to the first dose and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for 7 days prior to trial treatment.
7. Has an active autoimmune disease requiring systemic treatment within the past 3 months or a history of severe autoimmune disease or syndrome that requires steroids or immunosuppressive agents.
8. Has interstitial lung disease or active, non-infectious pneumonitis.
9. Has an active infection requiring systemic therapy.
10. Has a history or current evidence of any condition, therapy, or lab abnormality that might confound the results, interfere with the subject's participation, or is not in the best interest of the subject to participate, in the opinion of the investigator.
11. Has known psychiatric or substance abuse disorders that would interfere with the requirements of the trial.
12. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial.
13. Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2 treatment.
14. Has a history of HIV.
15. Has active Hepatitis B or Hepatitis C
16. Has received a live vaccine within 30 days prior to first dose.
17. Is currently being treated with ipilimumab (defined as ipilimumab < 6 weeks before first dose of treatment).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-01; Primary Completion 2018-06-08 (Actual); Study Completion 2018-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John M Richart, MD, Principal Investigator — Saint Louis University, Dept. of Internal Medicine, Div. of Hematology and Oncology
Locations (1):
- Saint Louis University Hospital, St Louis, Missouri, United States

REFERENCES:
- [Background] Ollila DW, Gleisner AL, Hsueh EC. Rationale for complete metastasectomy in patients with stage IV metastatic melanoma. J Surg Oncol. 2011 Sep;104(4):420-4. doi: 10.1002/jso.21961. PMID 21858837
- [Background] Laks S, Brueske KA, Hsueh EC. Neoadjuvant treatment of melanoma: case reports and review. Exp Hematol Oncol. 2013 Nov 8;2(1):30. doi: 10.1186/2162-3619-2-30. PMID 24499550
- [Background] Howard JH, Thompson JF, Mozzillo N, Nieweg OE, Hoekstra HJ, Roses DF, Sondak VK, Reintgen DS, Kashani-Sabet M, Karakousis CP, Coventry BJ, Kraybill WG, Smithers BM, Elashoff R, Stern SL, Cochran AJ, Faries MB, Morton DL. Metastasectomy for distant metastatic melanoma: analysis of data from the first Multicenter Selective Lymphadenectomy Trial (MSLT-I). Ann Surg Oncol. 2012 Aug;19(8):2547-55. doi: 10.1245/s10434-012-2398-z. Epub 2012 May 31. PMID 22648554
- [Background] Hamid O, Robert C, Daud A, Hodi FS, Hwu WJ, Kefford R, Wolchok JD, Hersey P, Joseph RW, Weber JS, Dronca R, Gangadhar TC, Patnaik A, Zarour H, Joshua AM, Gergich K, Elassaiss-Schaap J, Algazi A, Mateus C, Boasberg P, Tumeh PC, Chmielowski B, Ebbinghaus SW, Li XN, Kang SP, Ribas A. Safety and tumor responses with lambrolizumab (anti-PD-1) in melanoma. N Engl J Med. 2013 Jul 11;369(2):134-44. doi: 10.1056/NEJMoa1305133. Epub 2013 Jun 2. PMID 23724846

RESULTS

PARTICIPANT FLOW:
Groups:
- Pembrolizumab: Open-label non-randomized trial. All subjects will receive active drug (pembrolizumab).
  Assess the efficacy of neoadjuvant pembrolizumab in improving resectability rates in subjects with unresectable Stage III or unresectable Stage IV melanoma. Patients are eligible for study entry if complete metastectomy would be possible if the burden of disease can be decreased in size by up to 50%.
  Pembrolizumab: subjects will receive pembrolizumab, 200 mg infusions, every 3 weeks. Eligible subjects will receive at least 24 weeks of therapy and may receive up to 2 years of pembrolizumab therapy depending on response to treatment.
Period: Overall Study
Arm/Group | Pembrolizumab
Started | 10
Completed | 8
Not Completed | 2
Not completed — Lack of Efficacy | 2

BASELINE CHARACTERISTICS:
Groups:
- Pembrolizumab: Open-label non-randomized trial. All subjects will receive active drug (pembrolizumab).
  Pembrolizumab: subjects will receive pembrolizumab, 200 mg infusions, every 3 weeks. Eligible subjects will receive at least 24 weeks of therapy and may receive up to 2 years of pembrolizumab therapy depending on response to treatment.
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 10
Age, Continuous [Mean (Full Range); unit: years] | 66.3 [47 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Resectability Rate
Description: 'Resectability rate' is defined as the proportion of subjects in the trial that were unresectable at baseline who after treatment with pembrolizumab are now eligible for curative resection with complete metastectomy. The primary endpoint "resectability rate" is merely a novel statistical approach; it has no bearing on the duration of treatment that an individual patient may receive during the trial.
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 10
Participants
  Resectable | 8
  Unresectable | 2

2. Secondary Outcome: Response
Description: Response to treatment
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 10
Participants
  Complete Response | 1
  Resectable Partial Response | 7
  Resectable Progression of Disease | 1
  Progression of Disease | 1

ADVERSE EVENTS:
Time Frame: 24 months or: Subjects who meet all of the following criteria may discontinue follow up prior to 24 months: 1. CR or rPR with complete metastectomy has been confirmed. 2. Patient has received at least 24 weeks (8 cycles) of pembrolizumab therapy. 3. Patient has received at least 2 cycles of pembrolizumab after CR or rPR with complete metastectomy is documented.
Arm/Group | Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 3/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab (N=10)
Chest Pain (Cardiac disorders) | 1 (1)
Deep Vein Thrombosis (Blood and lymphatic system disorders) | 1 (1)
Hypophysitis (Endocrine disorders) | 1 (1)
Sclerosing Mesenteritis (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab (N=10)
Abdominal Pain (Gastrointestinal disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Headache (Nervous system disorders) | 4 (4)
Dizzy (Nervous system disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 3 (3)
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Folliculitis (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4)
Arm Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Neuropathy (Nervous system disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Leg Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Early Satiety (Gastrointestinal disorders) | 1 (1)
Vision Changes (Eye disorders) | 1 (1)
Postoperative Pain (Injury, poisoning and procedural complications) | 3 (3)
Hypertension (Vascular disorders) | 2 (2)
cyst (Skin and subcutaneous tissue disorders) | 1 (1)
Abrasion (Skin and subcutaneous tissue disorders) | 2 (2)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Postoperative Edema (Injury, poisoning and procedural complications) | 1 (1)
Postoperative Erythema (Injury, poisoning and procedural complications) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 1 (1)
Aspartate Aminotransferase Increased (Investigations) | 1 (1)
Alkaline Phosphatase Increased (Investigations) | 1 (1)
Sinus Infection (Infections and infestations) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Tooth Pain (Gastrointestinal disorders) | 1 (1)
Nocturia (Renal and urinary disorders) | 2 (2)
Weak Grip (Musculoskeletal and connective tissue disorders) | 2 (3)
Edema Axilla (General disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Foot Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Peripheral Edema (General disorders) | 2 (2)
Fatigue (General disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)
Thumb Cramp (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle Strain (Musculoskeletal and connective tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Limitations: a small number, 10 subjects, 9 of whom were male, participating in a study performed at a single institution.

Caveat: there was a disproportionate number of subjects with cutaneous disease only, i. e. no visceral metastases.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-08): https://cdn.clinicaltrials.gov/large-docs/50/NCT02306850/Prot_SAP_000.pdf